CLINICAL TRIAL: NCT01747980
Title: An Exploratory, Open-label Study to Evaluate the Safety of PRX-112 and Pharmacokinetics of Oral prGCD (Plant Recombinant Human Glucocerebrosidase) in Gaucher Patients
Brief Title: Safety and Pharmacokinetics of Oral PRX-112 in Gaucher Disease Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Protalix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB-112-01
Record Dates: First submitted 2012-12-05; First posted 2012-12-12 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Gaucher Disease
Keywords: Gaucher disease; human glucocerebrosidase; plant recombinant human glucocerebrosidase
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PRX-112 (Experimental): 250 mL of resuspended carrot cells administered orally in a vehicle
  Interventions: Drug: PRX-112

INTERVENTIONS:
Drug: PRX-112 — Single dose level, four doses per cohort
  Other Names: plant expressed recombinant human glucocerebrosidase

SUMMARY:
Absorption of therapeutic proteins taken orally has remained the major hurdle for treatment in humans. The proteins are generally degraded by enzymes in the stomach and intestine and the intestine lining that prevents absorption into the circulation. Administration of PRX-112, a plant recombinant human glucocerebrosidase (prGCD) using plant cells as carrier vehicle, may help overcome many of these hurdles. The plant cell wall protects the protein from degradation in its transport through the upper GI and allows release in the lower intestine. Studies in animals have shown that prGCD delivered in this way can be found in the blood stream in an active form.

DETAILED DESCRIPTION:
This exploratory, open-label safety and pharmacokinetic (PK) study is designed to assess the delivery of prGCD after oral administration of PRX-112 in Gaucher subjects. Subjects will receive an oral dose of PRX-112 in a single administration and followed by 3 consecutive daily administrations at the same dose. prGCD levels in plasma will be determined at selected time points. Safety parameters will also be assessed at selected time points. Enrollment will proceed into the next dosage cohort after the pharmacokinetic and safety data of the previous cohort have been reviewed. A different dosage may be selected based on the pharmacokinetic results of the first cohort.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years or older.
* Historical diagnosis of Gaucher disease with leukocyte GCD activity level ≤3 nmol/mg*hr (≤30 % of the mean activity of the reference range)
* Subjects who have not received enzyme replacement therapy (ERT) or substrate replacement therapy (SRT) in the past or patients who have not received ERT in the past twelve months
* Body Mass Index (BMI) 19 to 25 kg/m2 (inclusive).
* Non-smoking (by declaration) for a period of at least 6 months prior to screening visit.
* Subjects in generally good health in the opinion of the investigator as determined by medical history, vital signs and a physical examination.
* Negative hepatitis B or hepatitis C serology tests at screening.
* Ability to provide a written informed consent
* Female subjects of child-bearing potential or male subjects with female partners of child-bearing potential must agree to use two methods of contraception, one of which must be a barrier method. Acceptable methods of contraception include hormonal products, intrauterine device, or male or female condoms.

Exclusion Criteria:

* Presence of any co-morbidity other than Gaucher Disease
* Presence of any GIT disease or symptomatology suspected to be GIT related using a study specific GI questionnaire
* Subjects with any history of allergic response to drugs or other allergies deemed clinically significant or exclusionary for the study, including known food allergies
* History of alcohol or drug abuse
* Subjects who donated blood in the three months, or received blood or plasma derivatives in the six months, preceding study drug administration.
* Use of any investigational drug at screening or within 3 months of dosing.
* Subjects with an inability to communicate well with the investigators and study staff (i.e., language problem, poor mental development or impaired cerebral function).
* Subjects who are non-cooperative or unwilling to sign the consent form.
* Pregnant or nursing or planning to be pregnant during the study period.
* Have used any medication (excluding paracetamol), within 7 days of study drug administration including laxatives or other drugs, teas or food additives known to be used to treat constipation or diarrhea.
* Presence of any medical, emotional, behavioral or psychological condition that in the judgment of the investigator would interfere with the subject's compliance with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 3 days after the last dose
  Spontaneous reports of adverse events, or events identified during physical examination or clinical laboratory testing

SECONDARY OUTCOMES:
Area Under the Curve (AUC) | From start of infusion to 30 hours after infusion
  Area under the GCD level curve 0-30 hours (AUC0-30h)
Maximum Concentration (Cmax) | From start of infusion to 30 hours after infusion
Time of maximum prGCD concentration (Tmax) | From start of infusion to 30 hours after infusion

CONTACTS AND LOCATIONS:
Overall Officials: Einat Almon, PhD, Study Chair — Protalix Ltd.
Locations (2):
- Israel (2):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem